CLINICAL TRIAL: NCT00017368
Title: A Pilot Study Of Tandem High Dose Chemotherapy With Stem Cell Rescue Following Induction Therapy In Children With High Risk Neuroblastoma
Brief Title: Combination Chemotherapy Plus Peripheral Stem Cell Transplantation in Treating Children With Newly Diagnosed Neuroblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANBL00P1; COG-ANBL00P1 (Other: Children's Oncology Group); CDR0000068681 (Other: Clinical Trials.gov)
Record Dates: First submitted 2001-06-06; First posted 2003-10-09 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-02

CONDITIONS: Neuroblastoma
Keywords: regional neuroblastoma; disseminated neuroblastoma; localized unresectable neuroblastoma; stage 4S neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Filgrastim; sargramostim; Carboplatin; Cisplatin; Cyclophosphamide; Doxorubicin; Etoposide; etoposide phosphate; Ifosfamide; Isotretinoin; Melphalan; Thiotepa; Vincristine; Peripheral Blood Stem Cell Transplantation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All Patients (Experimental)
  Interventions: Biological: filgrastim; Biological: sargramostim; Drug: carboplatin; Drug: cisplatin; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: etoposide phosphate; Drug: ifosfamide; Drug: isotretinoin; Drug: melphalan; Drug: thiotepa; Drug: vincristine sulfate; Procedure: conventional surgery; Procedure: peripheral blood stem cell transplantation; Radiation: radiation therapy

INTERVENTIONS:
Biological: filgrastim
Biological: sargramostim
Drug: carboplatin
Drug: cisplatin
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: etoposide phosphate
Drug: ifosfamide
Drug: isotretinoin
Drug: melphalan
Drug: thiotepa
Drug: vincristine sulfate
Procedure: conventional surgery
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. Peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy followed by peripheral stem cell transplantation in treating children who have newly diagnosed neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxicity and feasibility of high-dose thiotepa and cyclophosphamide with autologous peripheral blood stem cell (PBSC) transplantation and sargramostim (GM-CSF) followed by high-dose carboplatin, etoposide, and melphalan with second PBSC transplantation, GM-CSF, and isotretinoin after induction in children with newly diagnosed high-risk neuroblastoma.
* Determine the role of the meta-iodobenzylguanidine (MIBG) scan in assessing response to tandem transplantation and minimal residual disease therapy in these patients.
* Determine the feasibility of quantitative polymerase chain reaction for neuroblastoma-specific ribonucleic acids at specific stages of treatment as a prognostic indicator of outcome in these patients.
* Determine the immune recovery by quantitation of lymphocyte subsets in these patients and limited functional analysis after completion of this regimen.

OUTLINE: This is a multicenter study. Patients are stratified according to peripheral blood stem cell (PBSC) selection (selected PBSCs vs unselected PBSCs). (Selected PBSC stratum closed to accrual as of 7/17/02.)

* Induction/harvest:

  * Course 1: Patients receive etoposide (VP-16) IV over 1 hour on days 2-4, cisplatin IV over 6 hours (beginning after VP-16 infusion) on days 1-5, and filgrastim (G-CSF) subcutaneously (SC) beginning on day 6 and continuing until blood counts recover.
  * Course 2: Patients receive vincristine IV and doxorubicin IV over 15 minutes on day 1, cyclophosphamide IV over 6 hours on days 1 and 2, and sargramostim (GM-CSF) SC beginning on day 3 and continuing until PBSC are harvested. Beginning after completion of course 2 and when blood counts recover, autologous PBSC are harvested.
  * Course 3: Patients receive VP-16 IV over 1 hour and ifosfamide IV over 1 hour on days 1-5 and G-CSF SC beginning on day 6 and continuing until blood counts recover.
  * Course 4: Patients receive VP-16 IV over 1 hour on days 1-3, carboplatin IV over 2 hours (beginning after VP-16 infusion) on days 1 and 2, and G-CSF SC beginning on day 4 and continuing until blood counts recover.
  * Course 5: Patients receive treatment as in course 2 but supported by G-CSF. Courses 1-5 each last 3-4 weeks. Patients undergo resection of the primary tumor after course 4 or 5 unless primary resection was completed at diagnosis (which is not recommended), no primary site is found, or the primary site is unresectable. Patients complete courses 1-5 and then proceed to the first conditioning/PBSC transplantation (PBSCT) in the absence of disease progression or unacceptable toxicity.
* First conditioning/PBSCT: Patients receive high-dose thiotepa IV on days -7 to -5 and cyclophosphamide IV over 1 hour on days -5 to -2. CD34+ PBSC are reinfused on day 0. GM-CSF is administered SC beginning on day 5 and continuing until blood counts recover. If blood counts have not recovered by day 28, unselected PBSC are reinfused. In the absence of disease progression or unacceptable toxicity, patients proceed to the second conditioning/PBSCT.
* Second conditioning/PBSCT: Beginning within 6-8 weeks after initiating the first conditioning, patients receive high-dose carboplatin IV continuously and etoposide phosphate IV continuously on days -7 to -4 and melphalan IV on days -7 to -5. PBSC and GM-CSF are administered as in the first PBSCT.

Beginning no earlier than day 28 after the second PBSCT, patients undergo local radiotherapy to the primary site and sites that are positive by meta-iodobenzylguanidine scan after induction twice a day for 7 days (or once a day for 12 days if twice daily dosing is not possible). Beginning on day 90 after the second PBSCT, patients receive oral isotretinoin twice a day for 2 weeks. Treatment repeats every 4 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 1 year, every 6 months for 1 year, and then annually thereafter.

PROJECTED ACCRUAL: A total of 31-39 patients will be accrued for this study within 22 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed high-risk neuroblastoma

  * Histologically proven AND/OR
  * Bone marrow specimen showing clumps of tumor cells accompanied by elevated urinary catecholamines
  * Age 1-30:

    * Must meet one of the following INSS staging criteria:

      * Stage IV regardless of biologic factors
      * Stage IIa/IIb with MYCN oncogene amplification (greater than 10) and unfavorable pathology
      * Stage III with MYCN oncogene amplification (greater than 10) or unfavorable pathology
      * Initially stage I, II, or IVS, that has progressed without interval chemotherapy
  * Under age 1:

    * INSS stage III, IV, or IVS with MYCN amplification (greater than 10)
* Must enter neuroblastoma biology study COG-ANBL00B1 within 2 weeks of diagnosis and before entry on this study

PATIENT CHARACTERISTICS:

Age:

* 30 and under at original diagnosis

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* No more than 1 prior course of chemotherapy on the intergroup low- or intermediate-risk neuroblastoma studies prior to determination of MYCN status and Shimada histology

Endocrine therapy:

* Not specified

Radiotherapy:

* Prior emergent radiotherapy to sites of function- or life-threatening neuroblastoma allowed

Surgery:

* Not specified

Other:

* No other prior systemic therapy for neuroblastoma

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2001-04; Primary Completion 2005-09 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Transplant-related mortality
  The endpoint used for early stopping rule 9.51 will be transplant-related mortality (TRM). A TRM is defined as any death occurring within 30 days after either the first or second HDC/SCR. The acceptable TRM rate is 7.5%. This rate is based on TRM rates previously observed in the prior CCG study 594, CCG study 3891, and POG study 9640 of 7%, 6%, and 0%, respectively.

SECONDARY OUTCOMES:
Incidence of symptomatic CMV, disseminated adenovirus infection, or EBV-LPD
  The endpoint to be used in assessing early stopping rule 9.52 will be the incidence of symptomatic CMV, disseminated adenovirus infection, or EBV-LPD. Patients with positive CMV antigenemia or CMV urine culture only (without symptoms of CMV infection), or patients who have a positive culture for adenovirus without evidence of dissemination, or patients with a positive EBV PCR who do not exhibit significant clinical signs (such as adenopathy) or symptoms will not trigger the stopping rule.
Event-free Survival | 1 year
  Assessment of feasibility and toxicity at the end of the study is time to event. Time to event is defined as the time from registration on the study until the first of the following events occurs: relapse, progression, secondary malignancy, or death, including toxic death. If none of those events occurs, then the time of last contact with the patient is used. Time to event will be used to calculate the one-year Event-free Survival (EFS) rate.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan A. Grupp, MD, PhD, Study Chair — Children's Hospital of Philadelphia
Locations (9):
- United States (8):
  - AFLAC Cancer Center and Blood Disorders Service of Children's Healthcare of Atlanta - Scottish RiteCampus, Atlanta, Georgia
  - Floating Hospital for Children, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia

REFERENCES:
- [Background] Marcus KJ, Shamberger R, Litman H, von Allmen D, Grupp SA, Nancarrow CM, Goldwein J, Grier HE, Diller L. Primary tumor control in patients with stage 3/4 unfavorable neuroblastoma treated with tandem double autologous stem cell transplants. J Pediatr Hematol Oncol. 2003 Dec;25(12):934-40. doi: 10.1097/00043426-200312000-00005. PMID 14663275
- [Background] Kletzel M, Katzenstein HM, Haut PR, Yu AL, Morgan E, Reynolds M, Geissler G, Marymount MH, Liu D, Kalapurakal JA, Shore RM, Bardo DM, Schmoldt J, Rademaker AW, Cohn SL. Treatment of high-risk neuroblastoma with triple-tandem high-dose therapy and stem-cell rescue: results of the Chicago Pilot II Study. J Clin Oncol. 2002 May 1;20(9):2284-92. doi: 10.1200/JCO.2002.06.060. PMID 11980999
- [Background] Donovan J, Temel J, Zuckerman A, Gribben J, Fang J, Pierson G, Ross A, Diller L, Grupp SA. CD34 selection as a stem cell purging strategy for neuroblastoma: preclinical and clinical studies. Med Pediatr Oncol. 2000 Dec;35(6):677-82. doi: 10.1002/1096-911x(20001201)35:63.0.co;2-h. PMID 11107145
- [Background] Grupp SA, Stern JW, Bunin N, Nancarrow C, Adams R, Gorlin JB, Griffin G, Diller L. Rapid-sequence tandem transplant for children with high-risk neuroblastoma. Med Pediatr Oncol. 2000 Dec;35(6):696-700. doi: 10.1002/1096-911x(20001201)35:63.0.co;2-0. PMID 11107149
- [Background] Grupp SA, Stern JW, Bunin N, Nancarrow C, Ross AA, Mogul M, Adams R, Grier HE, Gorlin JB, Shamberger R, Marcus K, Neuberg D, Weinstein HJ, Diller L. Tandem high-dose therapy in rapid sequence for children with high-risk neuroblastoma. J Clin Oncol. 2000 Jul;18(13):2567-75. doi: 10.1200/JCO.2000.18.13.2567. PMID 10893288